CLINICAL TRIAL: NCT05242328
Title: Comparison of Surgical Thoracoscopic Intercostal Nerve Block and Ultrasound-guided Erector Spinae Plane Block for Postoperative Analgesia and Enhanced Recovery After Uniportal Video-assisted Thoracoscopic Surgery: a Double-blinded, Randomized Controlled Trial
Brief Title: Postoperative Analgesia y After Uniportal Video-assisted Thoracoscopic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A-ER-110-293
Record Dates: First submitted 2022-01-26; First posted 2022-02-16 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2022-12

CONDITIONS: Post-operative Pain, Acute; Post-operative Pain; Thoracic Diseases; Post-Op Complication
Keywords: Uniportal video-assisted thoracoscopic surgery; Ultrasound-guided erector spinae plane block; surgical thoracoscopic intercostal nerve block; cumulative intravenous morphine consumption; visual analogue scale; Enhanced Recovery After Surgery
MeSH Terms: conditions — Pain, Postoperative; Thoracic Diseases; Postoperative Complications

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- post-operative VAS score of Ultrasound-guided erector spinae plane block (Active Comparator)
  Interventions: Procedure: Ultrasound-guided erector spinae plane block
- post-operative VAS score of surgical thoracoscopic intercostal nerve block (Active Comparator)
  Interventions: Procedure: surgical thoracoscopic intercostal nerve block

INTERVENTIONS:
Procedure: Ultrasound-guided erector spinae plane block — Ultrasound-guided erector spinae plane block
  Arms: post-operative VAS score of Ultrasound-guided erector spinae plane block
Procedure: surgical thoracoscopic intercostal nerve block — surgical thoracoscopic intercostal nerve block
  Arms: post-operative VAS score of surgical thoracoscopic intercostal nerve block

SUMMARY:
Ultrasound-guided erector spinae plane block (ESPB) is an interfascial blockade during thoracic anesthesia, first described by Forero in 2016, and is highlighted by technically feasibility and less complication rate. The patient is placed as decubitus position. The anesthesiologists use echo to identify the ipsilateral transverse process at T5 level, and insert the needle to 2-3 cm lateral to the spinous process until contact the transverse process. Then the injected local anesthetic will penetrate via erector spinae muscle to paravertebral space to affect and relieve pain.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, over 20 years old, u
* undergoing elective uniportal VATS lobectomy.

Exclusion Criteria:

* patient refusal,
* body mass index > 35 kg/m2,
* American society of anesthesiologists (ASA) grade above 3,
* contraindication to nerve block,
* allergy to analgesic agents,
* regular opioid used for chronic pain prior to this time surgery,
* conversion to thoracotomy or VATS procedure,
* postoperative intubation,
* postoperative intensive care unit admission.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-01-05 (Actual); Primary Completion 2024-12-26 (Estimated); Study Completion 2024-12-26 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scale | post-op 2 days
  post-op VAS score, 0-10, the higher means painful, and "0" point no pain.
accumulated morphine usage dose | post-op 2 days
  accumulated morphine usage dose

CONTACTS AND LOCATIONS:
Overall Officials: Shuoying Dai, Study Chair — National Cheng-Kung University Hospital
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan